CLINICAL TRIAL: NCT04599088
Title: Investigation of Brain Mechanisms Involved in the Urinary Continence Mechanism Associated With Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Becky Clarkson, Research Assistant Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20080217; R01AG065288 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Urgency Urinary Incontinence
Keywords: Urinary Incontinence; Urgency urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain functional MRI with simplified urodynamics (Experimental): Females with urgency urinary incontinence
  Interventions: Other: Brain functional MRI with simplified urodynamics

INTERVENTIONS:
Other: Brain functional MRI with simplified urodynamics — Structural:
  MPRAGE provides a structural image, which is used for coregistration of subjects. Structural scans are then performed including Diffusion Spectrum Imaging (DSI; microstructural), and Fluid-attenuated inversion recovery (FLAIR; white matter specific) scans.
  Functional:
  With about 50 ml in the bladder, resting state functional BOLD measurements are made, followed by functional whole-brain images while a small amount of saline is infused and withdrawn from the bladder, in 2 blocks of 4 repetitions each. Each repetition starts with a 12-scan pause, followed by infusion (6 scans = 12 s), pause (6 scans), and withdrawal (6 scans). Each block of 4 repetitions is completed by a 6 scan pause during which scanning continues. 24 ml is infused at 120 ml/min, and slightly less is withdrawn to avoid accommodation.This is repeated on an empty and full bladder along with a resting state image.

SUMMARY:
Urge urinary incontinence (UUI) is a common problem in older people which vastly reduces quality of life, yet the cause and mechanism of disease are not well understood. This study will characterize brain control of the bladder in young and old continent individuals and age-matched incontinent counterparts. This will expand the investigators current knowledge of how the brain controls the bladder, how that control changes with age and disease, and suggest new targets to guide development of better treatment.

DETAILED DESCRIPTION:
Current data suggest that bladder control comprises 3 cerebral circuits that maintain continence by suppressing the voiding reflex in the midbrain. In the UUI phenotype that responded to BFB (Biofeedback assisted pelvic floor muscle therapy), the mechanism involved enhancing deactivation of the first brain circuit (medial prefrontal cortex, mPFC) which resulted in less activation of the second circuit (which includes the midcingulate cortex). In the phenotype that was resistant to BFB, no brain changes were seen. Although the investigators have an emerging picture of the brain's role in UUI, the investigators have only rudimentary understanding of what is 'normal', i.e. how the brain normally controls the bladder. Moreover, the investigators do not know whether this control mechanism is the same across the lifespan, or whether it changes owing to the impact of aging. Thus, the investigators aims are to characterize the brain's normal role in bladder control in both young and old people, to determine the changes in brain structure and function that lead to bladder control failure (UUI), and to examine how such changes differ between young and old individuals. To address the aims, the investigators will utilize detailed neuroimaging to evaluate 80 asymptomatic women and 80 women with UUI, each group divided into young (18-45) and old (65+ years) individuals. The study will enable the investigators to define the brain's key structures, functional activity, and mechanisms involved in normal bladder control, and to identify the differences in these elements among those with UUI, both young and old.

By elucidating the mechanisms that mediate the brain's control (and loss of control) of bladder function, the proposed study should enhance the investigators working model, deepen the understanding of the impact of aging, and identify better targets for the treatment of UUI. It may thereby enable scientists to develop novel and more effective new therapies based on the revolution in neuroscience-and more hope for UUI sufferers.

ELIGIBILITY:
Inclusion Criteria:

* 'Old' (community-dwelling, mentally and functionally intact ambulatory women aged 65+ years) or 'Young' (equivalent women aged 18-45)
* 'Wet' (those who meet the International Continence Society definition of urgency urinary incontinence (urinary leakage accompanied by a sudden, strong urge to void which is difficult to defer) >5 times per week, for 3 months despite treatment for reversible causes (e.g., Urinary tract infection) and confirmed by a mean of one episode per day of UUI on 3-day bladder diary) or 'Dry' (women without current or past UUI or other lower urinary tract symptoms.) Infrequent stress incontinence of a small amount is acceptable.
* Urge-predominant mixed incontinence is acceptable provided the subject is able to differentiate between stress incontinence (SUI - leakage that coincides instantaneously with cough, laugh, exercise) and urgency incontinence, i.e., leakage accompanied by a sudden strong urge to void that is difficult to defer.
* Those with current or previous use of anticholinergic/beta-3 agonist medications will be considered for the study if they are willing to go through a washout period of at least 4 weeks of duration.

Exclusion Criteria:

Dry Groups

* Current or prior treatment for UUI
* Leakage on bladder diary not ascribed to minimal SUI (see bullet above)

All Groups: 'Wet' or 'Dry'; 'Young' or 'Old'

* Cognitive impairment:

  * MoCA<26
  * inability to perform a voiding diary/pad test
  * inability to reliably take daily medication
  * inability to comply with fMRI testing
* Impaired mobility

  o Timed up and go test ≥ 12 secs
* Medical instability:

  * severe uncontrolled hypertension >180mmHg systolic or >100mmHg diastolic
  * potential major changes in medical management over the course of the study period (i.e. upcoming surgery/treatment)
  * frailty according to the Fried criteria
* MRI incompatibility:

  * contraindicated metal implants
  * claustrophobia
  * unidentified/untested compatibility of metal implants
* Medication incompatibility:

  * allergy to study medication (all prophylactic antibiotic choices)
  * interaction of prophylactic antibiotic choices with current medications
  * expected change in medication during the study
* Neurological conditions:

  * spinal cord injury;
  * multiple sclerosis
  * clinically apparent lesions (e.g. lacunae associated with stroke)
  * prior stroke
  * Parkinson's Disease/ALS/MSA
  * any clinically apparent neurological condition
* Lower urinary tract comorbidities/treatment:

  * history of pelvic irradiation
  * bladder or advanced uterine cancer
  * possible urethral obstruction (advanced prolapse [POP-Q>II] or Qmax<12 ml/s on free flow)
  * urinary retention (PVR >200 ml)
  * Interstitial Cystitis/Bladder Pain Syndrome
  * artificial sphincter implant
  * Botox treatment for UUI within 1 year
  * Neuromodulation treatment for UUI
* Other comorbidities:

  * uncontrolled depression (PHQ-9 ≥10)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
BOLD (Blood oxygen level dependent) fMRI signal contrast | 20 minutes of a 1 hour MRI scan
  BOLD signal contrast - voxel-wise subtraction of normalized brain activity signal measure (BOLD response) during bladder fluid withdrawal from that during bladder infusion. Magnitude of BOLD contrast is then compared using ANOVA to compare the four groups (old dry/old wet/young dry/young wet). Differences are displayed as a map of t-values for each voxel of the brain, showing likelihood of statistical significance of differences. A priori regions of interest i.e. the bed nucleus of the stria terminalis (BST), pontine micturition center (PMC), periaqueductal grey (PAG), insula, medial prefrontal cortex (mPFC), dorsal anterior cingulate cortex/supplementary motor area (dACC/SMA) will be specified. Since BOLD signal represents the normalized contrast in fMRI signal between two states as a proxy for cerebral blood flow, it does not have a unit.

SECONDARY OUTCOMES:
Changes in brain structural integrity | 15 minutes of 1 hour MRI scan
  Difference in structural integrity of connective tracts will be compared using ANOVA to compare the four groups (old dry/old wet/young dry/young wet). Measure of structural integrity (normalized quantitative anisotropy, NQA), which describes the diffusion of water molecules around neuronal compartments (e.g., myelin, neurofilaments and microtubules) will be extracted from each individual and compared across groups.
Changes in brain structural integrity | 15 minutes of 1 hour MRI scan
  Difference in structural integrity of connective tracts will be compared using ANOVA to compare the four groups (old dry/old wet/young dry/young wet). Measure of structural integrity (generalized fractional anisotropy, GFA), which describes the diffusion of water molecules around neuronal compartments (e.g., myelin, neurofilaments and microtubules) will be extracted from each individual and compared across groups.
Functional connectivity during infusion/withdrawal task | 20 minutes of 1 hour MRI scan
  Functional connectivity calculated using generalized psychophysiological interaction (gPPI) analysis for each ROI (Eigenvariate time series; no units) will be extracted from the BOLD signal and a regression analysis performed, modeling the infusion/withdrawal blocks and the a priori ROI time series (mPFC, dACC/SMA, Insula) and its interactions with 'infuse' and 'withdraw' blocks.
Resting state analysis | 10 minutes of 1 hour MRI scan
  Resting state connectivity will be calculated by extracting the eigenvariate (no units) of three a priori selected ROIs (mPFC, dACC/SMA, Insula) and calculate voxel-wise connectivity maps for each region. Regional homogeneity evaluates regional changes in connectedness corresponding to local activation (temporal and spatial) between groups.
Differences in volume of brain structures | 10 minutes of 1 hour MRI scan
  Difference in grey matter volume (mm^3) on MRI as calculated by voxel based morphometry using ANOVA to compare the four groups (old dry/old wet/young dry/young wet). Grey matter volume of important brain structures will be compared.
Differences in white matter damage of brain structures | 10 minutes of 1 hour MRI scan
  Difference in volume of white matter damage (mm^3) on MRI using ANOVA to compare the four groups (old dry/old wet/young dry/young wet). Global volume of white matter damage will be compared. along with damage location.

CONTACTS AND LOCATIONS:
Overall Officials: Becky Clarkson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following publication, no end date
Access Criteria: Any purpose